CLINICAL TRIAL: NCT01211288
Title: Longitudinal Study of Dental Implant Therapy in HIV Positive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Toni Neumeier, Associate professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F090730003
Record Dates: First submitted 2010-09-28; First posted 2010-09-29 (Estimated); Results first posted 2020-05-15 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Dental Implant
Keywords: HIV; Implant; Crown

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- HIV negative group (Active Comparator): This group contains participants consented to receive implants and identified as negative for HIV
  Interventions: Device: Astra implants
- HIV positive group (Experimental): This group contains participants consented to receive implants and identified as positive for HIV
  Interventions: Device: Astra implants

INTERVENTIONS:
Device: Astra implants — Root form OsseoSpeed TX Astra Tech Implant System

SUMMARY:
The purpose is to place implants in HIV positive and HIV negative patients then follow patients over 3 years period of time to evaluate how well dental implants perform in HIV positive patients versus HIV negative patients.

DETAILED DESCRIPTION:
This study will review the osseointegration of implant supported restorations in HIV positive and HIV negative patients, then follow patients over a 3 year period of time. The treatment outcome as measured according to Mish criteria for implant success. Patients will be examined at each interval for the presence of pain, infection, mobility, and radiographic bone height of each implant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy enough to undergo the proposed therapy without compromise to existing health status
* At least 19 years old
* Able to read and understand written English without the aid of ad hoc interpretation
* Able to cognitively understand the proposed study and therapy and possible prognoses
* Able to consent for their own inclusion in the study.
* Implant supported restorations are limited to the following edentulous areas: Mandibular arch (excluding 2nd and 3rd molar areas), Maxillary anterior and premolar areas

Exclusion Criteria:

* Smoker
* Uncontrolled diabetes
* Uncontrolled hypertension
* Bisphosphonate user
* Bruxer
* Extraction site healed less than 6 months
* Women pregnant or lactating at the time of enrollment
* Previous malignant neoplasm
* A known hypersensitivity to Titanium metal
* Any medication/condition that in the opinion of the clinical investigators may adversely affect bone healing
* Any indication of an inability to make autonomous decisions

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-05 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toni T Neumeier, DMD, Principal Investigator — UAB Dental School
Locations (1):
- UAB Dental School, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To be determined

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HIV Negative Group | HIV Positive Group
Started | 21 | 20
Completed | 20 | 19
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Negative Group | HIV Positive Group | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 20 | 37
  >=65 years | 4 | 0 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 5 | 19
  Male | 7 | 15 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 11 | 12
  White | 12 | 9 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Implants Functioning in HIV Positive Subjects Compared to HIV Negative Subjects
Description: Dental implant supported restorations functioning in the mouth with no pain, no mobility, no infection and less than 50% bone loss around the implant site.
Time Frame: Baseline to 12 months after implant restoration complete
Population: Unable to do follow up on 3 participants - two participants from HIV negative group and one participant from HIV positive group, and one implant failure from HIV positive group
Measure: Number; unit: implants
Units Other Than Participants: implants
Arm/Group | HIV Negative Group | HIV Positive Group
Number analyzed (Participants) | 19 | 19
Number analyzed (implants) | 28 | 26
implants | 28 | 25

2. Primary Outcome: Number of Implants Functioning in HIV Positive Subjects Compared to HIV Negative Subjects
Description: Dental Implant supported restoration functioning in the mouth with no pain, no mobility, no infection and less than 50% bone loss around the implant site.
Time Frame: Baseline to 24 months after implant restoration complete
Population: Unable to do follow up on 7 participants, three participants from HIV negative group and four participants from HIV positive group
Measure: Number; unit: implants
Units Other Than Participants: implants
Arm/Group | HIV Negative Group | HIV Positive Group
Number analyzed (Participants) | 18 | 16
Number analyzed (implants) | 27 | 20
implants | 27 | 20

3. Primary Outcome: Number of Implants Functioning in HIV Positive Subjects Compared to HIV Negative Subjects
Description: as for outcome 2
Time Frame: Baseline to 36 months after implant restoration complete
Population: Unable to do follow up on 11 participants, five participants from HIV negative group and six participants from HIV positive group
Measure: Number; unit: implants
Units Other Than Participants: implants
Arm/Group | HIV Negative Group | HIV Positive Group
Number analyzed (Participants) | 16 | 14
Number analyzed (implants) | 25 | 17
implants | 25 | 17

4. Secondary Outcome: Peri-implant Health and Bone Maintenance as Measured by Radiographic Examination in HIV Positive Subjects Compared to HIV Negative Subjects
Description: Radiographic examination of implant osseointegration and bone loss by using traditional periapical and/or bitewing radiographs.
Time Frame: 12 months after implant restoration
Population: Unable to do follow up on three participants, two from HIV negative group and one from HIV positive group
Measure: Mean (Standard Deviation); unit: millmeters
Units Other Than Participants: implants
Groups:
- HIV Negative Group: This group contains participants consented to receive implants and identified as negative for HIV. Some participants has more than one implant.
  Astra implants: Root form OsseoSpeed TX Astra Tech Implant System
- HIV Positive Group: This group contains participants consented to receive implants and identified as positive for HIV.Some participants has more than one implant.
  Astra implants: Root form OsseoSpeed TX Astra Tech Implant System
Arm/Group | HIV Negative Group | HIV Positive Group
Number analyzed (Participants) | 19 | 19
Number analyzed (implants) | 28 | 25
millmeters | 0.34 (0.58) | 0.35 (0.71)

5. Secondary Outcome: Peri-implant Health and Bone Maintenance as Measured by Radiographic Examination in HIV Positive Subjects Compared to HIV Negative Subjects
Description: as for outcome 4
Time Frame: 24 months after implant restoration
Population: Unable to do follow up on 7 participants, three from HIV negative group and four from HIV positive group
Measure: Mean (Standard Deviation); unit: millmeters
Units Other Than Participants: implants
Arm/Group | HIV Negative Group | HIV Positive Group
Number analyzed (Participants) | 18 | 16
Number analyzed (implants) | 27 | 20
millmeters | 0.39 (0.49) | 0.33 (0.61)

6. Secondary Outcome: Peri-implant Health and Bone Maintenance as Measured by Radiographic Examination in HIV Positive Subjects Compared to HIV Negative Subjects
Description: Radiographic examination of implant osseointegration and bone loss by using traditional periapical and /or bitewing radiographs.
Time Frame: 36 months after implant restoration
Population: Unable to do follow up on 11 participants, five from HIV negative group and six from HIV positive group
Measure: Mean (Standard Deviation); unit: millmeters
Units Other Than Participants: implants
Arm/Group | HIV Negative Group | HIV Positive Group
Number analyzed (Participants) | 16 | 14
Number analyzed (implants) | 25 | 17
millmeters | 0.44 (0.52) | 0.48 (0.95)

ADVERSE EVENTS:
Time Frame: The specific period for this study was over 8 years from the time the first subject selected until 3 years follow up completed.
Description: Total 11 participants did not complete all follow up appointments through the end of the study. There are 5 in HIV negative group and 6 in HIV positive group.
Arm/Group | HIV Negative Group | HIV Positive Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

LIMITATIONS AND CAVEATS:
Based on a survey given every year, participants were extremely satisfied with the outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT01211288/Prot_SAP_000.pdf